CLINICAL TRIAL: NCT06699550
Title: The Effects of Haptonomy Application and Mindfulness-based Stress Reduction Program on Psychological Well-being Levels, Perceived Stress, and Fear of Childbirth in Primiparous Mothers: A Randomized Controlled Trial
Brief Title: Haptonomy and Mindfulness on Psychological Well-being Levels, Perceived Stress, Fear of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Asst. Prof, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-SBB-0435
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Mindfulness-Based Stress Reduction
Keywords: Primiparous women; Haptonomy; Mindfulness-based stress reduction program; Psychological well-being; Perceived stress; Fear of childbirth
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Haptonomy (Experimental): Haptonomy was conducted individually, both in a prenatal school and at home. At the beginning of the application, information was provided about the definition, purpose, and importance of haptonomy. It was stated that haptonomy would be carried out over 8 weeks, once a week for at least 30 minutes, on days and times of their choosing. In the first 4 weeks, it would be conducted under the guidance of the researchers, while in the following 4 weeks, it would be applied with the help of videos and brochures provided by the researchers, together with their partners.
  Interventions: Other: Haptonomy
- Mindfulness-Based Stress Reduction Program (Experimental): Participants were introduced to each other and provided with information related to pregnancy. The Mindfulness-Based Stress Reduction Program (MBSR) was introduced. The participants shared their levels of well-being, stress, coping mechanisms for fear of childbirth, and their expectations from the MBSR program. Awareness of habitual behaviors was facilitated. Afterwards, breath-focused meditation and dried fruit meditation were practiced. Participants were encouraged to maintain awareness of activities performed at any time during the day. Lastly, body scan meditation was taught, and participants were instructed to repeat the practice throughout the week using audio recordings sent via WhatsApp.
  Interventions: Other: Mindfulness-Based Stress Reduction Program
- Control (No Intervention): No use intervention.

INTERVENTIONS:
Other: Haptonomy — The session transitioned to energy work and dream visualization. The researcher and the pregnant participant placed their left hands on each other's hearts. The goal was for the participants to feel the energy flowing between them, sense their hearts, open their third eye, and prepare their hands. This exercise aimed to enhance the pregnant participant's confidence in her own emotions and body by recognizing her feelings and physical sensations. Next, the researcher and the pregnant participant placed their right hands on the participant's forehead and their left hands over their hearts. This positioning facilitated the pregnant participant in visually sensing the presence of her baby. It was intended to promote communication between the mother and her baby at both a physical and spiritual level.
  Arms: Haptonomy
Other: Mindfulness-Based Stress Reduction Program — Participants were introduced to each other and provided with information related to pregnancy. The Mindfulness-Based Stress Reduction Program (MBSR) was introduced. The participants shared their levels of well-being, stress, coping mechanisms for fear of childbirth, and their expectations from the MBSR program. Awareness of habitual behaviors was facilitated. Afterwards, breath-focused meditation and dried fruit meditation were practiced. Participants were encouraged to maintain awareness of activities performed at any time during the day. Lastly, body scan meditation was taught, and participants were instructed to repeat the practice throughout the week using audio recordings.
  Other Names: Mindfulness
  Arms: Mindfulness-Based Stress Reduction Program

SUMMARY:
Aim: The aim of this project was to examine the effects of haptonomy application and the mindfulness-based stress reduction program (MBSRP) on the psychological well-being levels, perceived stress, and fear of childbirth in primiparous women.

Materials and Methods: This prospective, single-blind, randomized controlled study was conducted between January 1, 2024, and October 1, 2024. A total of 120 primiparous women (40: control group, 40: haptonomy group, and 40: MBSRP group) who volunteered to participate in the study were randomly assigned to three groups: the intervention group (haptonomy and MBSRP) and the control group. The haptonomy and MBSRP groups received individual and face-to-face interventions for 8 weeks. At baseline, the 4th week, and the 8th week, the "Personal Data Collection Form," "Psychological Well-Being Scale," "Perceived Stress Scale," and "Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ/A) A version" were administered, based on a literature review.

ELIGIBILITY:
Inclusion Criteria:

* Women who are married and experiencing their first pregnancy.
* Aged 18 years or older.
* Able to read, write, and understand Turkish.
* Residing in the city center where the study is conducted.
* No physical or psychological health issues for themselves or their baby.
* Experiencing a spontaneous pregnancy between 22-28 weeks of gestation.
* Have not previously undergone BFTSAP (Body-Focused Therapy and Support for Anxiety during Pregnancy) and haptonomy applications.
* Pregnant women who agree to participate in the study.

Exclusion Criteria:

* Those with a known and diagnosed psychiatric disorder.
* Individuals who have previously undergone cognitive therapy.
* Experiencing severe levels of anxiety, stress, and depression.
* Having chronic diseases (such as hypertension, diabetes mellitus, heart diseases) that existed before or have emerged during pregnancy.
* Individuals who have not attended the first two sessions of the MBSR (Mindfulness-Based Stress Reduction) program and haptonomy applications.
* Lacking a partner or relative who can provide support and assistance at home during the applications.
* Without access to technical technology support.
* Pregnant women who do not agree to participate in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 40 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Psychological Well-Being Scale | change from starting to 4. and 8. week
  The Psychological Well-Being Scale, developed, consists of eight items aimed at measuring psychological well-being levels. The internal consistency coefficient of the scale is 0.87. The Turkish adaptation of the Psychological Well-Being Scale was conducted, who found the internal consistency coefficient to be 0.87 as well. The scale is rated on a 1-7 point scale, with higher scores indicating that the individual possesses psychological strengths.
Perceived Stress Scale | change from starting to 4. and 8. week
  The Perceived Stress Scale, consisting of 14 items, was developed to measure the degree to which individuals perceive certain situations in their lives as stressful. The scale is assessed using a 5-point Likert-type scoring system, ranging from 0 to 4. It comprises two factors: 'perception of stress/discomfort' and 'perception of inadequacy.' The scale allows for a maximum score of 56 and a minimum score of 0, with scores increasing as stress levels rise. The validity and reliability of the scale were established. The Turkish version of the Perceived Stress Scale (PSS-14) has an internal consistency coefficient of 0.84 and a test-retest reliability coefficient of 0.87.
Wijma Delivery Expectancy/Experience Scale (W-DEQ) Version A | change from starting to 4. and 8. week
  The scale, consists of 33 items. Responses to the items are rated on a scale from 0 to 5, utilizing a six-point Likert-type format. The maximum score attainable on the scale is 165, while the minimum is 0. A higher total score indicates a greater level of fear. Specifically, a scale score of 85 or above reflects clinical levels of birth fear, scores between 66 and 84 indicate severe fear, scores between 38 and 65 denote moderate fear, and scores of 37 and below signify mild levels of birth fear. The Cronbach's alpha coefficient for the scale is found to be 0.88 for first-time mothers (primiparous) and 0.90 for mothers who have given birth before (multiparous).

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided